CLINICAL TRIAL: NCT05682612
Title: Prognostic Value of Transcutaneous Partial Pressure of Oxygen in Patients With Novel Coronavirus Infection
Brief Title: Prognostic Value of PtcO2 in Patients With COVID-19
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Southeast University, China (Other)
Responsible Party: Principal Investigator, Jingyuan,Xu, Principal Investigator, Southeast University, China
Other Study IDs: 2023ZDSYLL001-P01
Record Dates: First submitted 2023-01-01; First posted 2023-01-12 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2023-10

CONDITIONS: COVID-19 Acute Respiratory Distress Syndrome
Keywords: ARDS; respiratory failure; COVID-19
MeSH Terms: conditions — Respiratory Insufficiency; COVID-19

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Survivors: Survivors of COVID-19 induced respiratory failure
  Interventions: Other: outcome; Other: Subtype of COVID-19
- Nonsurvivors: Nonsurvivors of COVID-19 induced respiratory failure
  Interventions: Other: outcome; Other: Subtype of COVID-19

INTERVENTIONS:
Other: outcome — hospital survivors and nonsurvivors
Other: Subtype of COVID-19 — Different subtype of COVID-19

SUMMARY:
Five percent of patients with COVID-19 progressed to respiratory failure and required ICU admission, such patients often have abnormal oxygen tolerance. However, there is still a lack of clinical indicators to predict the prognosis and treatment responsiveness of COVID-19.

DETAILED DESCRIPTION:
Five percent of patients with COVID-19 progressed to respiratory failure and required ICU admission. Attention should be paid to patients over 65 years of age who have severe underlying diseases (cancer, respiratory diseases, cardiovascular and cerebrovascular diseases, chronic renal failure, autoimmune deficiency diseases, etc.) and have not completed the whole course of vaccine, and such patients often have abnormal oxygen tolerance, that is, a significant decrease in skin finger pulse oxygen saturation (SpO2) can occur after daily activities. Basal SpO2 at admission is often associated with prognosis, but it is difficult to differentiate prognosis from responsiveness to treatment by changes in SpO2 after oxygen therapy is administered clinically. However, there is still a lack of clinical indicators to predict the prognosis and treatment responsiveness of COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-80 years, male or female; Patients with COVID-9 pneumonia (typical imaging features of COVID-19 pneumonia) (oxygen saturation ≤ 93% during air or arterial partial pressure of oxygen (PaO2)/oxygen concentration (FiO2) ≤ 300 mmHg at rest)；

Exclusion Criteria:

* Pregnant or lactating women; Patients who refuse to undergo transcutaneous tissue oxygen pressure monitoring; Clinicians believe that patients are not appropriate; Patients undergoing ECMO.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: COVID-19 patients
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2023-01-09 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Level of Transcutaneous partial pressure of oxygen | up to 30 days
  Level of Transcutaneous partial pressure of oxygen

SECONDARY OUTCOMES:
Level of Transcutaneous partial pressure of oxygen/FiO2 | up to 30 days
  Level of Transcutaneous partial pressure of oxygen/FiO2

CONTACTS AND LOCATIONS:
Overall Officials: Jingyuan Xu, M.D., Principal Investigator — Southeast University
Locations (1):
- Zhongda hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided